CLINICAL TRIAL: NCT04514328
Title: Highlighting the Benefits of Therapeutic Gardens in Alzheimer's Disease by 18F-FDG Cerebral PET /CT
Acronym: JAZTEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the study never opened for pandemic reasons
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: A202012345
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group (Experimental): patients with mild or moderate Alzheimer disease
  Interventions: Device: cerebral 18F-FDG PET-CT

INTERVENTIONS:
Device: cerebral 18F-FDG PET-CT — cerebral 18F-FDG PET-CT exam after walking in the garden while 2 weeks (75 minutes/per day from Monday to Friday)

SUMMARY:
The Alzheimer's Plan 2008-2012 allowed the installation of therapeutic gardens for the structures welcoming patients with Alzheimer's disease (AD) . The physical, psychological and social benefits are the improvement of the state of health and overall well-being.

There is a positive role in social interactions for patients with AD who can walk in the therapeutic gardens. Indeed, this promotes meetings with caregives and other people.

Using the garden decreases the stress level in patients (Ulrich). The therapeutic garden named "art, memory and life" in NANCY is based on art, nature and regional culture.

This garden can break with the "artificial" framework of care services often perceived as stressful.

In the garden, people walk around and have an experience that could improve self-image perception.

A clinical study with 2 groups of AD patients hospitalized in UCC or Cognitive Behavioral Unit took place in Nancy. The evaluation of the QCS (questionnaire on self-awareness) was carried out at the beginning and at the end of the study,

* a group of patients went into the garden: the QCS score increased
* a group of patients did not go to the garden (they remained in UCC): the QCS score decreased

ELIGIBILITY:
Inclusion Criteria:

* Patient with AD in the mild to moderate stage, followed at the memory and resource center (CMRR) (MMS 15-23) and having had a 18F-FDG PET-CT (Positon emission tomography) scan in routine care having a companion for the duration of the study .
* Patient with a neuropsychological assessment (MOCA, DO80, BREF, HAD) of less than 3 months. (If the last neuropsychological assessment dates from more than 3 months, these tests are carried out in routine care during the consultation was proposed and the consent obtained)
* Symptomatic treatment of AD (anticholinesterase or memantine) if prescribed, at a stable dose for 1 month, stable psychotropic treatment for 1 month
* Person affiliated with a social security scheme or beneficiary of such a scheme.
* Patient over 18 years old.
* Person received complete information on the organization of the research and having signed their informed consent.

Exclusion Criteria:

* Patient who did not have biomarkers identified by lumbar puncture
* Patient unable to perform a cerebral 18F-FDG PET-CT scan (lying position for more than 20 minutes)
* Patient unable to follow the therapeutic program of the garden.
* Woman of childbearing age whitout effective contraception.
* Pregnant woman or nursing mother.
* Person referred to in articles L. 1121-5, L. 1121-7 and L1121-8 of the public health code.
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric treatment under articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-02 (Estimated); Primary Completion 2022-10-06 (Estimated); Study Completion 2023-01-02 (Estimated)

PRIMARY OUTCOMES:
cerebral 18F-FDG PET-CT exam | up 20 days
  Topography of brain regions, whose carbohydrate metabolism has significantly changed in cerebral PET / CT with 18F-FDG before and after using the Therapeutic Garden.

SECONDARY OUTCOMES:
cerebral 18F-FDG PET-CT exam | up 20 days
  Topography of the brain regions, the carbohydrate metabolism of which has been significantly modified in cerebral PET / CT with 18F-FDG before and after the use of the therapeutic garden by people living with Alzheimer's disease by integrating the actimetry as co-variable in the model.
Comparison of QCS before and after using the therapeutic garden | up 18 days
  QCS is a self-awareness survey to be asked to patients before and after using garden
cerebral 18F-FDG PET-CT exam with QCS | up 20 days
  Topography of brain regions, whose carbohydrate metabolism covariates with clinical variables (QCS).
Modifications of the score of the electrodermal response during the use of the garden | up 14 days
  Electrodermal response is measured with sensors placed on the skin
cerebral 18F-FDG PET-CT exam with neuropsychological assessment | up 20 days
  Topography of brain regions, whose carbohydrate metabolism covariates with clinical neuropsychological assessment